CLINICAL TRIAL: NCT02796872
Title: The Effect of Feeding Infant Formula With Bimuno Galactooligosaccharide (GOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clasado (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CLA12016CN
Record Dates: First submitted 2016-05-30; First posted 2016-06-13 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-02

CONDITIONS: Dietary Modification

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- mother's breast milk. (Placebo Comparator): mother's breast milk.
  Interventions: Dietary Supplement: Mother's breast milk
- other GOS (Active Comparator): Commercial infant formula containing 4% w/w FOS:GOS (1:3)
  Interventions: Dietary Supplement: GOS
- B-GOS 3% (Experimental): Commercial infant formula containing 3% w/w FOS:B -GOS (1:2)
  Interventions: Dietary Supplement: B-GOS 3%
- B-GOS 2% (Experimental): Commercial infant formula containing 4% w/w FOS:B -GOS (1:3)
  Interventions: Dietary Supplement: B-GOS 2%

INTERVENTIONS:
Dietary Supplement: GOS — GOS resource (β-galactosidase from Bacillus circulans) Commercial infant formula containing 4% w/w FOS:GOS (1:3)
  Arms: other GOS
Dietary Supplement: B-GOS 3% — Bimuno-GOS (B-GOS) resource (β-galactosidase from Bifidobacteriumbifidum) Commercial infant formula containing 3% w/w FOS:B -GOS (1:2)
  Arms: B-GOS 3%
Dietary Supplement: B-GOS 2% — Bimuno-GOS (B-GOS) resource (β-galactosidase from Bifidobacteriumbifidum) Commercial infant formula containing 4% w/w FOS:B -GOS (1:3)
  Arms: B-GOS 2%
Dietary Supplement: Mother's breast milk — exclusively breastfed infants for at least 7 days prior to enrollment
  Arms: mother's breast milk.

SUMMARY:
This survey is a multicenter, double-blind, randomized, controlled, parallel-designed, prospective trial and is intended to evaluate the Bimuno GOS effects on growth, tolerance, gut health, fecal flora and immune function.

ELIGIBILITY:
Inclusion Criteria:

* o 15 ± 3 days of age at randomization, inclusive (day of birth is considered day 0)

  * Singleton birth
  * Gestational age of 37-42 weeks (36 weeks and six days is considered 36 weeks gestational age)
  * Birth weight of 2500g to 4000g
  * Signed informed consent obtained for infant's participation in the survey
  * Parent or guardian of infant agrees not to enroll infant in another interventional clinical research survey while participating in this survey
  * APGAR score after 5 minutes of life > 7
  * Consuming only one source of nutrition
  * Formula-fed infant: Infant consuming infant formula as the sole source of nutrition for 7 consecutive days prior to randomization
  * Breastfed infant: Infant consuming mother's breast milk as the sole source of nutrition for 7 consecutive days prior to registration

Exclusion Criteria:

* Infant with inborn malformation and with hereditary and/or chronic and/or inborn diseases requiring hospital care superior to 7 days
* Diseases jeopardizing intrauterine growth
* Weight at Visit 1 is <95% of birth weight [(weight at Visit 1÷birth weight) x 100 <95%]
* Infant born from mother suffering from metabolic and/or chronic diseases
* Infant with an acute infection or gastroenteritis at time of randomization or registration
* Infant consuming supplemental foods
* Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake at time of randomization or registration
* Infant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as Combined Immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich Syndrome, Severe Congenital Neutropenia and Secondary Immunodeficiencies linked to HIV infection, Down Syndrome or others) and children with known head/brain disease/injury such as Microcephaly, Macrocephaly or others

Ages: 12 Days to 18 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 392 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Anthropometric parameters | 6 months
  body length, body weight, and head circumferences at enrollment (15± 3 days of age), 30, 60, 90, 120, 150 and 180 days of age
Fecal bacteria analysis | 6 months
  o Fecal bacteria analysis of Bifidobacterium, Lactobacillus, Clostridium perfringens and Escherichia coli at the enrollment 30 days of age ,120 days of age and 180 days of age

SECONDARY OUTCOMES:
Dietary | 6 months
  tool characteristics, tolerance, formula acceptance, stress and 3-day well-being (quality of life) questionnaire prior to each survey visit recorded at 30, 60, 90, 120, 150 and 180 days of age
Formula intake | 6 months
  Formula intake (24-hour dietary recall) at 30, 60, 90, 120, 150 and 180 days of age
All medically confirmed adverse events and antibiotic record | 6 months
  All medically confirmed adverse events including crying, gaseous colics, regurgitation, vomit, skin rashes, fever and concomitant medications recorded on medical records as a measure of safety and tolerability throughout the survey period.
Fecal sIgA and SCFA analysis | 6 months
  Fecal sIgA and SCFA analysis at 30 days of age (visit 1) and 180 days of age (visit 6)
Saliva cortisol, IgA, chromogranin A and lysozyme | 6 months
  Saliva cortisol, IgA, chromogranin A and lysozyme at 30, 90 and 180 days of age